CLINICAL TRIAL: NCT00607347
Title: Atenolol Exposure as Risk for Adverse Metabolic Responses to Beta Blockers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UF IRB 591-2007; U01GM074492 (NIH); GCRC grant RR00082
Record Dates: First submitted 2008-01-15; First posted 2008-02-05 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension
Keywords: Keywords by National Institute of General Medical Sciences; Hypertension; Adverse metabolic effects; Beta blockers; Dyslipidemia; Atenolol; New onset diabetes; Pharmacokinetic study; Oral glucose tolerance test
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): The subjects will be undergoing a oral glucose tolerance test.
  Interventions: Other: Glucose

INTERVENTIONS:
Other: Glucose — Oral Glucose Tolerance Test

SUMMARY:
The researchers hypothesize that the impact of increasing systemic exposure to atenolol leads to increased risk for adverse metabolic effects from atenolol therapy in hypertension. This will be accomplished through a 24-hour pharmacokinetic (PK) study and oral glucose tolerance test in hypertensive patients taking chronic atenolol 100 mg daily.

DETAILED DESCRIPTION:
The current study is a sub-study of Pharmacogenomic Evaluation of Antihypertensive Responses (PEAR - NCT00246519). The primary objective of this pharmacokinetic (PK) study is to investigate the correlation of atenolol Cp with hypertriglyceridemia and insulin sensitivity in mild to moderate hypertensive patients after 6-8 weeks of atenolol treatment.

Participants will undergo the PK study when they have been on atenolol 100 mg once daily for at least 4 weeks and on atenolol therapy (50 mg or 100 mg) for ≥ 7 weeks. They will undergo a two hour Oral Glucose Tolerance Test (OGTT), 1 hour after atenolol dosing. Blood will be drawn at 12 time points for 24 hours. Atenolol Cp will be measured in all 12 blood samples and will be correlated with the glucose/insulin measured during the OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from PEAR who are on atenolol 100 mg once daily will be invited to participate
* Other inclusion criteria from PEAR

Exclusion Criteria:

* Patients with BMI >35 kg/m2 will be excluded
* Other exclusion criteria from PEAR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Correlation of area under curve (AUC) up to 24 hour time point of atenolol plasma drug concentrations and glucose/insulin values obtained from OGTT and triglycerides | Glucose/insulin will be measured during 2 hour Oral Glucose Tolerance Test and from baseline measurements from PEAR, triglycerides will be measured from baseline lab measurements from PEAR and during the pharmacokinetic study

SECONDARY OUTCOMES:
HDL-cholesterol, fatty acids, total cholesterol | Baseline lab values from PEAR and before the start of pharmacokinetic study

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Johnson, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States